CLINICAL TRIAL: NCT02482090
Title: T Cell Therapy for Patients With Metastatic Ovarian Cancer
Brief Title: TIL Therapy for Metastatic Ovarian Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Inge Marie Svane (Other)
Responsible Party: Sponsor-Investigator, Inge Marie Svane, M.D., Professor, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GY1508
Record Dates: First submitted 2015-06-23; First posted 2015-06-25 (Estimated); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Metastatic Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Cyclophosphamide; fludarabine; fludarabine phosphate; Interleukin-2; aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patient group (Experimental): All patients receive the same treatment. Alle patients are hospitalized during treatment (approximately 3 weeks) and receive treatment only once.
  Stem Cells are harvested a minimum of 3 weeks before treatment for potential later use if the patients are having difficulties recovering from the lymphodepleting chemotherapy.
  The patients are admitted to hospital day -8 and receive lymphodepleting chemotherapy (cyclophosphamide and fludarabine= on day -7 to day -1.
  The TILs are infused on day 0 and Interleukin-2 therapy is administered on day 0 to day 5.
  Interleukin-2 is administered in an i.v. continous decrescendo regimen starting approximately 6 hours after TIL infusion with a duration of approximately 5 days.
  Stem Cells can be administered after treatment if needed.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Biological: TIL infusion; Drug: Interleukin-2

INTERVENTIONS:
Drug: Cyclophosphamide — Cyclophosphamide 60 mg/kg is administered i.v. on day -7 and day -6.
  Other Names: Cyclophospamide
Drug: Fludarabine — Fludarabine 25 mg/m2 is administered on day -5 to day -1.
  Other Names: Fludarabinephosphate; Fludara
Biological: TIL infusion — The maximum number of expanded TILs are infused over 30-45 minutes on day 0.
  Other Names: T Cell infusion
Drug: Interleukin-2 — Interleukin-2 is administered as a continous i.v. infusion in a decrescendo regimen (18 MIU/m3 IL-2 over 6 hours, 18 MIU/m2 IL-2 over 12 hours, 18 MIU/m2 IL-2 over 24 hours followed by 4,5 MIU/m2 IL-2 over another 24 hours for three days).
  Other Names: IL-2; Proleukin

SUMMARY:
Adoptive T cell therapy with tumor infiltrating lymphocytes (TIL) has achieved impressive clinical results with durable complete responses in patients with metastatic melanoma. The TILs are isolated from patients own tumor tissue followed by in vitro expansion and activation for around 4-6 weeks. Before TIL infusion the patients receive 1 week of preconditioning chemotherapy with cyclophosphamide and fludarabine. After TIL infusion Interleukin-2 is administered to support T cell acitivation and proliferation in vivo.

Recent studies suggest, that TIL therapy works in other cancers than Metastatic Melanoma, including Ovarian Cancer. In this study TIL therapy is administered to patients with metastatic Ovarian Cancer.

DETAILED DESCRIPTION:
Adoptive T cell therapy with tumor infiltrating lymphocytes (TIL) has achieved impressive clinical results with durable complete responses in patients with metastatic melanoma. The TILs are isolated from patients own tumor tissue followed by in vitro expansion and activation for around 4-6 weeks. Before TIL infusion the patients receive 1 week of preconditioning chemotherapy with cyclophosphamide and fludarabine. After TIL infusion Interleukin-2 is administered to support T cell acitivation and proliferation in vivo.

Objectives:

To evaluate safety and feasibility when treating patients with metastatic ovarian cancer with ACT with TILs.

To evaluate treatment related immune responses To evaluate clinical efficacy

Design:

Patients will be screened with a physical exam, medical history, blood samples and ECG.

Patients will undergo surgery to harvest tumor material for TIL production. Patients is admitted day -8 in order to undergo lymphodepleting chemotherapy with cyclophosphamide and fludara starting day -7.

On day 0 patients receive TIL infusion and shortly after starts IL-2 infusion continually following the decrescendo regimen.

The patients will followed until progression or up to 5 years

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed high grade serous adenokarcinoma ovarian cancer metastasis available for surgical resection (more than 1 cm3) and residual measurable disease after resection
* Progression/reccurence of ovarian cancer after 1. line platin based chemotherapy or progression/reccurence after 2. line or additional chemotherapy
* ECOG performance status 0-1
* Life expectancy > 6 months
* No significant toxicity from prior treatments, except sensoric- and motoric neuropathia and/or alopecia
* Adequate renal, hepatic and hematological function
* Women of childbearing potentil (WOCBP) must be using an effective method of contraception during treatment and for at least 6 months after completion of treatment
* Able to comprehend the information given and willing to sign informed consent

Exclusion Criteria:

* Other malignancies, unless followed for ≥ 5 years with no sign of disease
* Severe allergies, history of anaphylaxis or known allergies to the administered drugs.
* Serious medical or psychiatric comorbidity
* Creatinine clearance < 70 ml/min
* Acute or chronic infection with e.g. HIV, hepatitis, tuberculosis
* Severe and active autoimmune disease
* Pregnant and nursing women
* Need for immunosuppressive treatment, e.g. corticosteroids or methotrexate
* Concomitant treatment with other experimental drugs
* Patients with uncontrolled hypercalcemia
* Less than four weeks since prior systemic antineoplastic treatment at the time of treatment

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-07; Primary Completion 2016-12 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Number and type of reported adverse events | 0-24 weeks
  Determine the safety of the administration of TIL therapy including lymphodepleting chemotherapy and Interleukin-2 for patients with metastatic Ovarian Cancer by reporting adverse events according to CTCAE v. 4.0.

SECONDARY OUTCOMES:
Treatment related immune responses | Up to 12 months
  To evaluate the immunological impact of TIL therapy for patients with metastatic Ovarian Cancer
Objective response rate | Up to 12 months
  Clinical responses will be evaluated by RECIST 1.1.
Overall Survival | Up to 12 months
  Overall Survival (OS), defined as time from treatment initiation to death, will be described with use of Kaplan Meier curve.
Progression free survival | Up to 12 months
  Progression free survival (PFS), defined as the time from treatment initiation to disease progression, relapse or death due to any cause, which ever comes first, will be described with Kaplan Meier curve.

CONTACTS AND LOCATIONS:
Overall Officials: Inge Marie Svane, Prof., MD, Study Director — Center for Cancer Immune Therapy, Dept of Hematology/Oncology, Copenhagen University Hospital Herlev, Herlev Ringvej 75, DK-2730; Magnus Pedersen, MD, Principal Investigator — Center for Cancer Immune Therapy, Dept of Hematology/Oncology, Copenhagen University Hospital Herlev, Herlev Ringvej 75, DK-2730
Locations (1):
- Center for Cancer Immune Therapy Dept. of Hematology/oncology, Copenhagen, Herlev, Denmark

REFERENCES:
- [Derived] Westergaard MCW, Andersen R, Chong C, Kjeldsen JW, Pedersen M, Friese C, Hasselager T, Lajer H, Coukos G, Bassani-Sternberg M, Donia M, Svane IM. Tumour-reactive T cell subsets in the microenvironment of ovarian cancer. Br J Cancer. 2019 Feb;120(4):424-434. doi: 10.1038/s41416-019-0384-y. Epub 2019 Feb 5. PMID 30718808
- [Derived] Andersen R, Donia M, Westergaard MC, Pedersen M, Hansen M, Svane IM. Tumor infiltrating lymphocyte therapy for ovarian cancer and renal cell carcinoma. Hum Vaccin Immunother. 2015;11(12):2790-5. doi: 10.1080/21645515.2015.1075106. PMID 26308285